CLINICAL TRIAL: NCT04614506
Title: Transcranial Magnetic Stimulation to Measure Cortical Excitability in Dravet Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Encoded Therapeutics (Industry)
Responsible Party: Principal Investigator, Alexander Rotenberg, Associate, Department of Neurology; Director, Neuromodulation Program; Associate Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Other Study IDs: IRB-P00034206
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Transcranial Magnetic Stimulation; Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject with DS: Participants will complete two visits spaced out by 4 - 8 weeks to undergo neurophysiological assessments (Electroencephalogram [EEG], and Transcranial magnetic stimulation [TMS]).
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Electroencephalogram (EEG)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation (TMS) is a method for noninvasive electrical cortical stimulation, where small intracranial currents are generated by a powerful, fluctuating, extracranial magnetic field. TMS is unique in its capacity for experimental, diagnostic, and therapeutic utility. Single pulse (spTMS) and paired-pulse TMS (ppTMS) have been used extensively to study, measure, and modulate cortical excitability and plasticity.
  Other Names: Nexstim Navigated Brain Stimulation (NBS) System 4
Device: Electroencephalogram (EEG) — These will be an ambulatory EEG recordings that span 24 hours and done without sedation. Recordings will be performed using electrode locations specified by the international 10-20 system for standard clinical practice.
  Other Names: Natus

SUMMARY:
Dravet syndrome (DS) is an epileptic encephalopathy caused by pathogenic variants in the SCN1A gene resulting in medically refractory epilepsy and psychomotor delays.

As a pilot study assessing for feasibility, the investigators aim to test whether alterations in cortical excitatory:inhibitory ratio can be reliably recorded. The investigators will utilize transcranial magnetic stimulation (TMS) metrics of cortical excitatory and inhibitory tone as an initial step towards translating findings from rodent genetic models of DS into disease-specific biomarkers and offer future measures of therapeutic target engagement in this patient population.

Participants will complete two visits, each consisting of a TMS session and an EEG session. Visits will be scheduled 4-8 weeks apart.

DETAILED DESCRIPTION:
This is a single site study to be conducted at Boston Children's Hospital (BCH) investigating the neurophysiological biomarkers of epilepsy and developmental disability in children and young adults with Dravet Syndrome.

Mechanistically, the features of the DS phenotype are attributable to a loss of cortical inhibition. TMS is a non-invasive form of focal cortical stimulation in which an external powerful magnet induces an electrical field intracranially over the stimulated region that is used to interrogate or modulate states of cortical excitation or inhibition.

Accordingly, the investigators propose to test whether metrics of cortical excitability and inhibition can be obtained by transcranial magnetic stimulation (TMS) and EEG in patients with DS.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months - 30 years
* Ability to obtain informed consent with the participant or legally authorized representative
* DS confirmed by pathogenic variant in SCN1A gene
* Medical history consistent with clinical phenotype of DS

Exclusion Criteria:

* Comorbid conditions such as a second genetic diagnosis which may confound interpretation.
* Current or planned participation in a clinical drug or device trial.
* Previous participation in a gene therapy or gene editing trial
* Allergy to adhesives used for surface EMG electrodes
* Contraindications to TMS (e.g. implanted devices for which there is no TMS safety data)

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adults diagnosed with Dravet Syndrome.
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Resting motor threshold (% machine output) | 1 year
  Resting motor threshold (rMT) is obtained by single-pulse TMS and measures voltage-gated sodium-channel-mediated cortical excitability. It is the minimum intensity of stimulation needed to reliably evoke a motor evoked potential (MEP) of at least 50 microvolts in over 50% of trials. It is reported as a percentage of total machine output.
Durations of cortical silent period (ms) | 1 year
  Cortical Silent Period (CSP) is a single-pulse TMS measure of GABA-mediated cortical inhibition, in which stimulation is applied to the motor cortex while subjects are activating a target muscle (here, abductor pollicis brevis and deltoid muscles), resulting in a pause in muscle contraction. The time between stimulation and the return of voluntary muscle activity is the CSP, measured in milliseconds (ms).
Ratio of motor evoked potential amplitudes (no units) | 1 year
  Facilitation (ICF) are paired-pulse TMS metrics of cortical inhibition and excitability, respectively. A short interval interstimulus (1-5 ms) leads to cortical inhibition reflective of GABAergic neurotransmission; a longer interval interstimulus of 10-20 ms leads to a cortical facilitation, which reflects glutamatergic neurotransmission; an even longer interstimulus interval of 50-300 ms reflects GABAB-mediated local inhibition and likely GABAA-mediated network inhibition. The ratio of the peak-to-peak amplitude (in mm) of the second MEP to the first (or control) MEP will be calculated for each of these stimulation protocols.
Cortical Inhibitory Tone | 1 year
  Power in the gamma (30-80 Hz) frequency band.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rotenberg, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No